CLINICAL TRIAL: NCT04050358
Title: The Effect of Basis™ and High Intensity Interval Training (HIIT) on Muscle Metabolism and Exercise Performance in Healthy 18 - 35 Year Olds
Brief Title: Effect of Basis™ and High Intensity Interval Training (HIIT) on Muscle Metabolism and Exercise Performance
Status: Withdrawn | Phase: Phase 1 | Type: Interventional
Why Stopped: Lack of Funds
Sponsor: Elysium Health (Industry)
Collaborators: University of Exeter (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Double | Purpose: Other
Other Study IDs: Basis-HIIT
Record Dates: First submitted 2019-08-06; First posted 2019-08-08 (Actual); Last update posted 2023-02-15 (Actual); Status verified 2023-02

CONDITIONS: Healthy

STUDY DESIGN:
Who Masked: Participant, Investigator
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No | US Export: Yes

ARMS (2):
- 1X dose of NRPT (Active Comparator)
  Interventions: Dietary Supplement: NRPT
- Placebo (Placebo Comparator)
  Interventions: Dietary Supplement: Placebo oral capsule

INTERVENTIONS:
Dietary Supplement: NRPT — Subjects randomly assigned to the active group will receive Nicotinamide Riboside and Pterostilbene (each capsule contains 125 mg NR and 25 mg PT, total daily dose is 2 capsules) for 3 weeks
  Other Names: BasisTM
  Arms: 1X dose of NRPT
Dietary Supplement: Placebo oral capsule — Subjects randomly assigned to the Placebo group will receive placebo oral capsules for 3 weeks
  Arms: Placebo

SUMMARY:
This is a single-center, randomized, placebo-controlled pilot study to evaluate the effects of high intensity interval training (HIIT) and daily administration of BasisTM for 3 weeks, in 18-35 year old males.

The study will consist of a screening visit, baseline visit, followed by treatment and HIIT phase (3 weeks) and a post-supplementation, follow-up visit (this will occur 48 h (or more) after the final HIIT session). Following the screening phase, subjects who meet entry criteria will be randomly assigned to 1 of 2 treatment groups: recommended dose of BasisTM (250 mg Nicotinamide Riboside and 50 mg Pterostilbene) per day or matching-placebo in a 1:1 ratio.

ELIGIBILITY:
Inclusion Criteria:

* 18 to 35 year old males
* Body mass index between 18.5-30 kg.m-2
* Ability to give informed consent
* Recreationally active (defined in the present study as exercising once a week or more).

Exclusion Criteria:

* Those regularly conducting HIIT or highly trained in endurance events (e.g. triathlete)
* Currently taking supplements known to affect metabolism (e.g. ibuprofen, stimulants, vitamins, NR)
* Taking prescribed medication
* Consuming a vegan diet
* Consuming a high fat, low carbohydrate diet
* Habitual consumption of protein and/or dairy supplements (e.g. whey protein)
* Smokers

Ages: 18 Years to 35 Years | Sex: Male | Healthy Volunteers: Yes
Age Groups: Adult
Enrollment: 0 (Actual)
Dates: Start 2023-02 (Estimated); Primary Completion 2023-04 (Estimated); Study Completion 2023-05 (Estimated)

PRIMARY OUTCOMES:
Mitochondrial function | 3 weeks
  Measured via high-resolution respirometry using the Oroboros Oxygraph

SECONDARY OUTCOMES:
Exercise Capacity | 3 weeks
  To measure maximal endurance capacity measured via VO2max
Muscle strength | 3 weeks
  To measure maximal voluntary contraction using a force transducer strength chair
Muscle power | 3 weeks
  Determine the effects of HIIT with and without NRPT supplementation on muscle power producing capabilities measured by the 30 second Wingate test
Mitochondrial proteins | 3 weeks
  To determine whether HIIT with NRPT supplementation improves mitochondrial function more so than HIIT alone, using Western blotting
Body Mass | 3 weeks
  To determine the effects of HIIT with and without NRPT supplementation on body composition by measuring body mass using a bioelectrical impedance analysis scale
Percent Body Fat | 3 weeks
  To determine the effects of HIIT with and without NRPT supplementation on body composition by measuring percent body fat using a bioelectrical impedance analysis scale
Recovery via POMS | 3 weeks
  To determine the effects of HIIT with and without NRPT supplementation on recovery via profile of mood states (POMS)
Recovery via RESTQ | 3 weeks
  To determine the effects of HIIT with and without NRPT supplementation on recovery via recovery stress (RESTQ) questionnaire
Physical activity levels using FitBit | 3 weeks
  To characterize volunteer's habitual physical activity levels.
Height | 3 weeks
  Measure height using a stadiometer, to characterize demographics of recruited volunteers the recruited volunteers
Blood pressure | 3 weeks
  Measure blood pressure using Dinamap Pro monitor to characterize demographics of recruited volunteers the recruited volunteers

CONTACTS AND LOCATIONS:
Overall Officials: Timothy Etheridge, PhD, Principal Investigator — University of Exeter
Locations (1):
- University of Exeter, Exeter, United Kingdom

IPD SHARING:
Plan to Share IPD: No